CLINICAL TRIAL: NCT03889860
Title: Objective Choroidal Thickness Measurements During Intraocular Inflammation in Uveitis Using Optical Coherence Tomography
Brief Title: Objective Choroidal Thickness Measurements in Uveitis
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Wroclaw Medical University (Other)
Collaborators: Wrocław University of Science and Technology (Other)
Responsible Party: Principal Investigator, Joanna Przeździecka-Dołyk, Principal Investigator, Wroclaw Medical University
Other Study IDs: ST-859 extention
Record Dates: First submitted 2019-03-23; First posted 2019-03-26 (Actual); Last update posted 2022-03-29 (Actual); Status verified 2022-03

CONDITIONS: Uveitis
MeSH Terms: conditions — Uveitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Uveitis group
- Control group: age and sex matched group to the uveitis group

SUMMARY:
Optical Coherence Tomography (OCT) machines are non-contact instruments that can provide micrometer scale imaging of biological tissue. Applying the image processing allows us to automatically measure the choroidal thickness with good interclass correlation coefficient to the manual measurements.

ELIGIBILITY:
Inclusion Criteria:

* To the control group - ability to perform OCT examination
* To the uveitis group - with one or more of the following clinical features (as indicators for active state of the disease):

  1. >1+ anterior chamber cells;
  2. >1+ vitreous haze;
  3. presence of vitreous cells;
  4. presence of blood in anterior chamber;
  5. presence of blood in vitreous;
  6. presence of aqueous or vitreous pigment.

Exclusion Criteria:

* To the control group - diagnosed uveitis
* In case of all groups:

  1. inability to give informed consent;
  2. inability to maintain stable fixation for OCT imaging.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Uveitis patients and matched control group
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2018-09-01 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Submacular choroidal thickness in different stages of the disease | 5 years
  OCT EDI recordings processed with developed by researchers methodology for image processing

SECONDARY OUTCOMES:
ETDRS Visual Acuity | 1 year
  Visual Acuity will be performed with ETDRS charts different for right and left eye
The SUN working group grading system for anterior chamber cells | 1 year
  At each visit anterior chamber will be examined to assess anterior chamber cells (1mm x 1mm slit beam in height and width, when thrown at an angle of 45-60°). The recorded number of cells will be used to determine the grade according to the SUN criteria.
The SUN working group grading system for anterior chamber flare | 1 year
  At each visit anterior chamber will be examined to assess anterior chamber flare (1mm x 1mm slit beam in height and width, when thrown at an angle of 45-60°). The observed changes will be used to determine the grade according to the SUN criteria.
AREDS 2008 Clinical Lens Opacity Grading Procedure | 1 year
  Using AREDS system for classifying cataracts from photographs: AREDS Report No. 4 the lens opacity will be graded
NIH grading system for vitreous cells | 1 year
  At each visit vitreous will be examined to assess vitreous cells (1mm x 3mm slit beam in anterior vitreous). The recorded number of cells will be used to determine the grade according to the NIH criteria.
NIH grading system for vitreous haze | 1 year
  At each visit vitreous will be examined to assess vitreous haze. The recorded of clarity of posterior pole funduscopy will be used to determine the grade according to the NIH criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Marta Misiuk-Hojło, Professor, Study Chair — Medical University of Wrocław
Locations (1):
- Department of Ophthalmology, Wroclaw, Poland

IPD SHARING:
Plan to Share IPD: Undecided
Intention to share anonymised data of each patient visit in the study

REFERENCES:
- [Background] Indaram M, Agron E, Clemons TE, Sperduto RD, Wong WT, Ferris FL 3rd, Chew EY; Age-Related Eye Disease Study Research Group. Changes in lens opacities on the age-related eye disease study grading scale predict progression to cataract surgery and vision loss: age-related eye disease study report no. 34. Ophthalmology. 2015 May;122(5):888-96. doi: 10.1016/j.ophtha.2014.12.037. Epub 2015 Feb 11. PMID 25682177
- [Background] Li Y, Lowder C, Zhang X, Huang D. Anterior chamber cell grading by optical coherence tomography. Invest Ophthalmol Vis Sci. 2013 Jan 9;54(1):258-65. doi: 10.1167/iovs.12-10477. PMID 23249705
- [Background] Passaglia CL, Arvaneh T, Greenberg E, Richards D, Madow B. Automated Method of Grading Vitreous Haze in Patients With Uveitis for Clinical Trials. Transl Vis Sci Technol. 2018 Mar 23;7(2):10. doi: 10.1167/tvst.7.2.10. eCollection 2018 Mar. PMID 29600118
- [Background] Davis JL, Madow B, Cornett J, Stratton R, Hess D, Porciatti V, Feuer WJ. Scale for photographic grading of vitreous haze in uveitis. Am J Ophthalmol. 2010 Nov;150(5):637-641.e1. doi: 10.1016/j.ajo.2010.05.036. Epub 2010 Aug 16. PMID 20719302
- [Background] Keane PA, Karampelas M, Sim DA, Sadda SR, Tufail A, Sen HN, Nussenblatt RB, Dick AD, Lee RW, Murray PI, Pavesio CE, Denniston AK. Objective measurement of vitreous inflammation using optical coherence tomography. Ophthalmology. 2014 Sep;121(9):1706-14. doi: 10.1016/j.ophtha.2014.03.006. Epub 2014 May 15. PMID 24835759
- [Background] Madow B, Galor A, Feuer WJ, Altaweel MM, Davis JL. Validation of a photographic vitreous haze grading technique for clinical trials in uveitis. Am J Ophthalmol. 2011 Aug;152(2):170-176.e1. doi: 10.1016/j.ajo.2011.01.058. Epub 2011 Jun 8. PMID 21652026